CLINICAL TRIAL: NCT00876148
Title: Risk of Hepatitis B Virus Reactivation in Patients Undergoing Allografting
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Other Study IDs: LAM Allo SCT
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Hepatitis B Virus; Allograft; Hematological Malignancies
Keywords: Incidence of hepatitis B after allografting; Risk of hepatitis B reactivation; Lamivudine prophylaxis
MeSH Terms: conditions — Hepatitis B; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to evaluate the risk of hepatitis B reactivation in patients undergoing allografting.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an allograft for hematological malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients undergoing allografting for hematological malignancies
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera S Giovanni Battista, Torino, Italy

REFERENCES:
- [Derived] Giaccone L, Festuccia M, Marengo A, Resta I, Sorasio R, Pittaluga F, Fiore F, Boccadoro M, Rizzetto M, Bruno B, Marzano A. Hepatitis B virus reactivation and efficacy of prophylaxis with lamivudine in patients undergoing allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2010 Jun;16(6):809-17. doi: 10.1016/j.bbmt.2009.12.533. Epub 2010 Jan 7. PMID 20060484